CLINICAL TRIAL: NCT03842176
Title: Clinical Application of CTC in Operable Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, ZHOU Yidong, Professor, Peking Union Medical College Hospital
Other Study IDs: PUMCH-BREAST-CTC
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; CTC; Neoadjuvant chemotherapy; Adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemotherapy: CTC of operable breast cancer patients with neoadjuvant chemotherapy before surgery in different periods: before neo-chemotherapy, during neo-chemotherapy, on surgery day, after surgery and follow-up time.
  Interventions: Procedure: Neoadjuvant chemotherapy before surgery
- Surgery: CTC of operable breast cancer patients with surgery followed by adjuvant chemotherapy in different periods: on surgery day, after surgery, before adjuvant chemotherapy, during adjuvant chemotherapy, and follow-up time.
  Interventions: Procedure: Surgery followed by adjuvant chemotherapy

INTERVENTIONS:
Procedure: Neoadjuvant chemotherapy before surgery — The operable breast cancer patients takes neoadjuvant chemotherapy before surgery.
  Groups: Neoadjuvant chemotherapy
Procedure: Surgery followed by adjuvant chemotherapy — The operable breast cancer patients takes surgery followed by adjuvant chemotherapy.
  Groups: Surgery

SUMMARY:
The investigators aim to evaluate the possibility of clinical application of CTC detection in samples or peripheral blood of breast cancer patients, so as to act as the new techniques or indicators of early diagnosis, therapy efficiency, or postoperative surveillance of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures.
* Age of at least 18 and at most 70 years.
* Performance status (Karnofsky-Index) >80%.
* Chemotherapy is necessary before or after surgery.
* No clinical evidence of local recurrence or distant metastases.
* Complete staging work-up within 3 months prior to registration. All patients must have (bilateral) mammography or breast MRI, chest X-ray; other tests may be performed as clinically indicated.
* Life expectancy of at least 2 years, disregarding the diagnosis of cancer.
* Adequate organ function including normal red and white blood count, platelets, serum creatinine, bilirubin, and transaminases within normal range of the institution.
* Patients must be available for and compliant to treatment and follow-up.
* Patients registered on this trial must be treated and followed up at the participating center.

Exclusion Criteria:

* Known hypersensitivity reaction to the investigational compounds or incorporated substances.
* Local recurrence and/or metastasis of breast cancer.
* No need of chemotherapy.
* Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration.
* Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix).
* Any other serious medical pathology, such as congestive heart failure; unstable angina; history of myocardial infarction during the previous year; uncontrolled high risk arrhythmias.
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study.
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operable breast cancer patients who need chemotherapy before or after surgery.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The level of CTC mRNA markers in patients' peripheral blood | 3 years
  The level of CTC mRNA markers in patients' peripheral blood of neoadjuvant chemotherapy group and surgery group in different periods

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China